CLINICAL TRIAL: NCT04799158
Title: A Phase 2, Randomized, Double-Blind, Multicenter Study to Evaluate the Efficacy and Safety of Vonoprazan 10 mg, 20 mg, and 40 mg Compared to Placebo for Relief of Episodic Heartburn in Subjects With Symptomatic Non-Erosive Gastroesophageal Reflux Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of Vonoprazan Compared to Placebo in Participants With Symptomatic Non-Erosive Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Phathom Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NERD-201
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Results first posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Non-Erosive Gastro-Esophageal Reflux Disease; Heartburn
Keywords: Symptomatic Non-Erosive Gastroesophageal Reflux Disease; NERD; Vonoprazan; Heartburn
MeSH Terms: conditions — Heartburn | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: During the Run-In Period, participants will receive open-label vonoprazan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Run-In Period (Experimental): Participants will receive vonoprazan 20 mg once daily for up to 4 weeks.
  Interventions: Drug: Vonoprazan
- Vonoprazan 10 mg: On-Demand Treatment Period (Experimental): Participants who have stable disease (no heartburn on the last 7 days of the Run-In Period) will take vonoprazan 10 mg when heartburn occurs during the 6 week On-Demand Treatment Period. Participants can take no more than one dose in a 24 hour period.
  Interventions: Drug: Vonoprazan
- Vonoprazan 20 mg: On-Demand Treatment Period (Experimental): Participants who have stable disease (no heartburn on the last 7 days of the Run-In Period) will take vonoprazan 20 mg when heartburn occurs during the 6 week On-Demand Treatment Period. Participants can take no more than one dose in a 24 hour period.
  Interventions: Drug: Vonoprazan
- Vonoprazan 40 mg: On-Demand Treatment Period (Experimental): Participants who have stable disease (no heartburn on the last 7 days of the Run-In Period) will take vonoprazan 40 mg when heartburn occurs during the 6 week On-Demand Treatment Period. Participants can take no more than one dose in a 24 hour period.
  Interventions: Drug: Vonoprazan
- Placebo: On-Demand Treatment Period (Placebo Comparator): Participants who have stable disease (no heartburn on the last 7 days of the Run-In Period) will take a placebo when heartburn occurs during the 6 week On-Demand Treatment Period. Participants can take no more than one dose in a 24 hour period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vonoprazan — Orally via capsules
  Arms: Run-In Period; Vonoprazan 10 mg: On-Demand Treatment Period; Vonoprazan 20 mg: On-Demand Treatment Period; Vonoprazan 40 mg: On-Demand Treatment Period
Drug: Placebo — Orally via capsules
  Arms: Placebo: On-Demand Treatment Period

SUMMARY:
The primary objectives of this study are to assess the efficacy of vonoprazan (10 mg, 20 mg, and 40 mg On-Demand) compared to placebo (On-Demand) in relief of episodic heartburn over 6 weeks in participants with symptomatic non-erosive gastroesophageal reflux disease (NERD), and to assess the safety of vonoprazan (10 mg, 20 mg, and 40 mg On-Demand) compared to placebo (On-Demand) in participants with symptomatic NERD.

ELIGIBILITY:
Inclusion Criteria for Run-In Period

1. The participant is ≥18 years of age at the time of informed consent signing.
2. In the opinion of the investigator or sub investigators, the participant is capable of understanding and complying with protocol requirements.
3. The participant signs and dates a written informed consent form (ICF) and any required privacy authorization prior to the initiation of any study procedures. The participant is informed of the full nature and purpose of the study, including possible risks and side effects. The participant has the ability to cooperate with the investigator. Ample time and opportunity should be given to read and understand verbal and/or written instructions.
4. The participant identified their main symptom as heartburn, a burning sensation in the retrosternal area (behind the breastbone).
5. History of episodes of heartburn for 6 months or longer prior to screening.
6. Heartburn reported on 4 or more days during any 7 consecutive days in the Screening Period as recorded in the electronic diary.
7. A female participant of childbearing potential who is or may be sexually active with a non sterilized male partner agrees to routinely use adequate contraception from the signing of informed consent until 4 weeks after the last dose of study drug.

Inclusion Criteria for On-Demand Treatment Period

1. The participant completes the Run-In Period, during which the participant was at least 80% compliant with open-label study drug.
2. The participant has stable disease, ie, no heartburn the last 7 days of the Run-In Period.
3. The participant continues to fulfill all eligibility criteria for the Run-In Period (except Inclusion Criteria 4).
4. Participant completes at least 80% of diary entries during Run-In Period, including 80% of diary entries over the last 7 days.

Exclusion Criteria for Run-In Period

1. Endoscopically confirmed erosive esophagitis (EE) during the Screening Period assessed by the investigator. Endoscopy should be performed after participants meet Inclusion Criteria 6. Any endoscopic confirmation performed in a routine clinical setting within 7 days before signing the informed consent is acceptable to use for the purpose of fulfilling the screening requirement.
2. The participant has active irritable bowel syndrome (IBS) or had a flare of IBS requiring therapy within the prior 6 months.
3. The participant has a history of or is suspected of having functional heartburn diagnosed by the Rome IV criteria.
4. The participant has a history of or is suspected of having functional dyspepsia diagnosed by the Rome IV criteria.
5. The participant has endoscopic Barrett's esophagus (>1 cm of columnar-lined esophagus) and/or definite dysplastic changes in the esophagus.
6. The participant has any other clinically significant condition affecting the esophagus, including eosinophilic esophagitis; esophageal varices; viral or fungal infection; esophageal stricture; a history of radiation therapy, radiofrequency ablation, endoscopic mucosal resection, or cryotherapy to the esophagus; or any history of caustic or physiochemical trauma (including sclerotherapy or esophageal variceal band ligation). However, participants diagnosed with Schatzki's ring (mucosal tissue ring around lower esophageal sphincter) or hiatal hernia are eligible to participate.
7. The participant has scleroderma (systemic sclerosis).
8. The participant has a history of surgery or endoscopic treatment affecting gastroesophageal reflux, including fundoplication and dilation for esophageal stricture (except Schatzki's ring) or a history of gastric or duodenal surgery (except endoscopic removal of benign polyps).
9. The participant has an active gastric or duodenal ulcer within 4 weeks before the first dose of study drug.
10. Use of prescription or non-prescription proton pump inhibitors (PPIs) or histamine-2 receptor antagonists (H2RAs) throughout the study.
11. The participant has received vonoprazan in a clinical trial at any time or any other investigational compound (including those in post-marketing studies) within 30 days prior to the start of the Screening Period. A participant who has been screen failed from another clinical study and who has not been dosed may be considered for enrollment in this study.
12. The participant is a study site employee, an immediate family member, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or who may have consented under duress.
13. The participant has cutaneous lupus erythematosus or systemic lupus erythematosus.
14. The participant has had clinically significant upper or lower gastrointestinal bleeding within 4 weeks prior to screening.
15. The participant has Zollinger-Ellison syndrome or other gastric acid hypersecretory conditions.
16. The participant has a history of hypersensitivity or allergies to vonoprazan (including the formulation excipients: D-mannitol, microcrystalline cellulose, hydroxypropyl cellulose, fumaric acid, croscarmellose sodium, magnesium stearate, hypromellose, macrogol 8000, titanium oxide, or red or yellow ferric oxide). Skin testing may be performed according to local standard practice to confirm hypersensitivity.
17. The participant has a history of alcohol abuse, illegal drug use, drug addiction, or regularly consumes >21 units of alcohol (1 unit = 12 oz/300 mL beer, 1.5 oz/25 mL hard liquor/spirits, or 5 oz/100 mL wine) per week based on self-report within the 12 months prior to screening. Participants must have a negative urine drug screen for cannabinoids/ tetrahydrocannabinol and nonprescribed medications at screening. Participants taking prescription drugs (except prescription cannabinoids/tetrahydrocannabinol) will be allowed.
18. The participant is taking any excluded medications or treatments listed in the protocol.
19. If female, the participant is pregnant, lactating, or intending to become pregnant before, during, or within 4 weeks after participating in this study, or intending to donate ova during such time period.
20. The participant has a history or clinical manifestations of significant central nervous system, cardiovascular, pulmonary, hepatic, renal, metabolic, other gastrointestinal, urological, endocrine, or hematological disease that, in the opinion of the investigator, would confound the study results or compromise participant safety.
21. The participant requires hospitalization or has surgery scheduled during the course of the study or has undergone major surgical procedures within 30 days prior to the Screening Visit.
22. The participant has a history of malignancy or has been treated for malignancy within 5 years prior to the start of the Screening Period (Visit 1). (The participant may be included in the study if he/she has recovered from cutaneous basal cell carcinoma or cervical carcinoma in situ).
23. The participant has acquired immune deficiency syndrome (AIDS) or human immunodeficiency virus (HIV) infection, or tests positive for the hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or HCV ribonucleic acid (HCV-RNA). However, participants who test positive for HCV antibody but negative for HCV-RNA are permitted to participate.
24. The participant has any of the following abnormal laboratory test values at the start of the Screening Period:

    1. Creatinine levels: >2 mg/dL (>177 μmol/L)
    2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 × the upper limit of normal (ULN) or total bilirubin >2 × ULN (except participants with Gilbert Syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2022-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Phathom Pharmaceuticals
Locations (63):
- United States (63):
  - Pinnacle Research Group, Anniston, Alabama
  - North Alabama Research Center LLC, Athens, Alabama
  - Medical Affiliated Research Center Inc, Huntsville, Alabama
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Del Sol Research Management - Clinedge, Tucson, Arizona
  - Preferred Research Partners - ClinEdge, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - GW Research, Inc, Chula Vista, California
  - eStudySite, Chula Vista, California
  - Paragon Rx Clinical, Garden Grove, California
  - OM Research LLC, Lancaster, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Paragon Rx Clinical, Inc., Santa Ana, California
  - Western States Clinical Research Inc, Wheat Ridge, Colorado
  - Imagine Research of Palm Beach County, Boynton Beach, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - ENCORE Borland-Groover Clinical Research, Jacksonville, Florida
  - ClinCloud, Maitland, Florida
  - G. Medical Center, Orlando, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Precision Clinical Research, LLC, Sunrise, Florida
  - Guardian Angel Research Center, Tampa, Florida
  - Florida Medical Clinic, LLC Clinical Research Division, Zephyrhills, Florida
  - IACT Health, Columbus, Georgia
  - In Quest Medical Research, Suwanee, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Care Access, Chicago, Illinois
  - Iowa Digestive Disease Center, Clive, Iowa
  - Clinical Trials Management LLC, Covington, Louisiana
  - Legacy Clinical Solutions: Tandem Clinical Research, LLC, Marrero, Louisiana
  - Clinical Trials Management LLC, Metairie, Louisiana
  - Investigative Clinical Research, Annapolis, Maryland
  - Gastroenterology Associates of Western Michigan, PLC, Wyoming, Michigan
  - GI Associates and Endoscopy Center, Flowood, Mississippi
  - Quality Clinical Research, Omaha, Nebraska
  - Sierra Clinical Research - ClinEdge, Las Vegas, Nevada
  - Site 2, Las Vegas, Nevada
  - Site 1, Las Vegas, Nevada
  - Advanced Research Institute, Reno, Nevada
  - Drug Trials America, Hartsdale, New York
  - Javara Inc, Charlotte, North Carolina
  - Medication Management LLC, Greensboro, North Carolina
  - Carolina Research, Greenville, North Carolina
  - Peters Medical Research, LLC, High Point, North Carolina
  - Trial Management Associates LLC, Wilmington, North Carolina
  - Remington Davis Inc, Columbus, Ohio
  - Frontier Clinical Research, LLC, Uniontown, Pennsylvania
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Rapid City Medical Center LLP, Rapid City, South Dakota
  - Clinical Research Associates Inc, Nashville, Tennessee
  - Inquest Clinical Research, Baytown, Texas
  - Family Medicine Associates of Texas, Carrollton, Texas
  - Synergy Group US, LLC, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Rio Grande Gastroenterology, McAllen, Texas
  - Quality Research Inc, San Antonio, Texas
  - Gastroenterology Research of San Antonio (GERSA), San Antonio, Texas
  - Sherman Clinical Research, Sherman, Texas
  - Advanced Research Institute, Ogden, Utah
  - Advanced Research Institute, Sandy City, Utah
  - Virginia Gastroenterology Institute, Suffolk, Virginia

IPD SHARING:
Plan to Share IPD: No
Data from this study will be published; however, it is undecided if patient level data will be made available at this time.

REFERENCES:
- [Derived] Fass R, Vaezi M, Sharma P, Yadlapati R, Hunt B, Harris T, Smith N, Leifke E, Armstrong D. Randomised clinical trial: Efficacy and safety of on-demand vonoprazan versus placebo for non-erosive reflux disease. Aliment Pharmacol Ther. 2023 Nov;58(10):1016-1027. doi: 10.1111/apt.17728. Epub 2023 Sep 26. PMID 37750406

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was performed at 54 sites in the United States between 25 March 2021 and 17 January 2022. Of the 1115 participants screened for the study, 458 participants were enrolled into the Run-In Period. Of these participants, 207 participants were randomized to receive study drug in the On-Demand treatment period.
Pre-assignment Details: Eligible participants who had symptomatic NERD were initially dosed during an open-label Run-In Period with vonoprazan 20 mg once per day (QD) for 4 weeks. Participants with stable disease (defined by those who had no heartburn on the last 7 consecutive days of the Run-In Period) and were compliant with the electronic diary and study drug were randomized using a 1:1:1:1 allocation ratio to receive either vonoprazan 10 mg, 20 mg, or 40 mg or placebo during the 6-week On-Demand Treatment Period.
Groups:
- Run-In Period: Participants received oral vonoprazan 20 mg once daily (QD) for up to 4 weeks.
- Vonoprazan 10 mg: On-Demand Treatment Period: Participants who had stable disease (no heartburn on the last 7 days of the Run-In Period) received oral vonoprazan 10 mg when heartburn occurred during the 6 week On-Demand Treatment Period. Participants could take no more than one dose in a 24-hour period.
- Vonoprazan 20 mg: On-Demand Treatment Period: Participants who had stable disease (no heartburn on the last 7 days of the Run-In Period) received oral vonoprazan 20 mg when heartburn occurred during the 6 week On-Demand Treatment Period. Participants could take no more than one dose in a 24-hour period.
- Vonoprazan 40 mg: On-Demand Treatment Period: Participants who had stable disease (no heartburn on the last 7 days of the Run-In Period) received oral vonoprazan 40 mg when heartburn occurred during the 6 week On-Demand Treatment Period. Participants could take no more than one dose in a 24-hour period.
- Placebo: On-Demand Treatment Period: Participants who had stable disease (no heartburn on the last 7 days of the Run-In Period) received oral placebo when heartburn occurred during the 6 week On-Demand Treatment Period. Participants could take no more than one dose in a 24-hour period.
Period: Run-In Period
Arm/Group | Run-In Period | Vonoprazan 10 mg: On-Demand Treatment Period | Vonoprazan 20 mg: On-Demand Treatment Period | Vonoprazan 40 mg: On-Demand Treatment Period | Placebo: On-Demand Treatment Period
Started | 458 | 0 | 0 | 0 | 0
Completed | 207 | 0 | 0 | 0 | 0
Not Completed | 251 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0 | 0 | 0
Not completed — Significant Protocol Deviation | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 0 | 0 | 0 | 0
Not completed — Miscellaneous | 3 | 0 | 0 | 0 | 0
Not completed — Did not meet On-Demand Eligibility Criteria | 226 | 0 | 0 | 0 | 0
Period: On-Demand Treatment Period
Arm/Group | Run-In Period | Vonoprazan 10 mg: On-Demand Treatment Period | Vonoprazan 20 mg: On-Demand Treatment Period | Vonoprazan 40 mg: On-Demand Treatment Period | Placebo: On-Demand Treatment Period
Started | 0 | 52 | 52 | 51 | 52
Completed | 0 | 51 | 52 | 49 | 48
Not Completed | 0 | 1 | 0 | 2 | 4
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Significant Protocol Deviation | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Miscellaneous | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: On-Demand Treatment Period: The Safety On-Demand Set included all participants in the Safety Run-In Set who were randomized and treated at least one heartburn episode with randomized treatment during the On-Demand Treatment period.
Groups:
- Placebo: On-Demand Treatment Period: Participants who had stable disease (no heartburn on the last 7 days of the Run-In Period) received oral placebo when heartburn occured during the 6 week On-Demand Treatment Period. Participants could take no more than one dose in a 24-hour period.
- Total: Total of all reporting groups
Arm/Group | Vonoprazan 10 mg: On-Demand Treatment Period | Vonoprazan 20 mg: On-Demand Treatment Period | Vonoprazan 40 mg: On-Demand Treatment Period | Placebo: On-Demand Treatment Period | Total
Number analyzed (Participants) | 49 | 49 | 48 | 47 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (11.89) | 55.7 (12.87) | 52.0 (14.60) | 52.7 (15.20) | 53.7 (13.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 33 | 25 | 33 | 118
  Male | 22 | 16 | 23 | 14 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 17 | 15 | 12 | 60
  Not Hispanic or Latino | 33 | 32 | 33 | 35 | 133
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 32 | 36 | 39 | 29 | 136
  Black or African-American | 7 | 5 | 6 | 10 | 28
  Asian | 8 | 6 | 3 | 7 | 24
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0
  Unknown | 1 | 0 | 0 | 0 | 1
  Not reported | 1 | 1 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Evaluable Heartburn Episodes Completely Relieved Within 3 Hours and With No Further Heartburn Reported for 24 Hours After Taking Study Drug
Description: An evaluable heartburn episode was an episode for which study drug was taken and for which the participant completed at least one entry in the heartburn episode diary.
  For a heartburn episode to be considered completely relieved, a participant must not have taken rescue antacid within 3 hours of taking study drug. For sustained relief, complete relief must have been accompanied by 24 hours without another heartburn episode after taking study drug.
Time Frame: On-Demand Treatment Period: Day 1 to Day 42
Population: Intent-to-Treat (ITT) On-Demand Set: includes all participants in the Safety Run-In set who were randomized and completed at least one heartburn episode diary during the On-Demand Treatment Period.
Measure: Number; unit: percentage of heartburn episodes
Units Other Than Participants: evaluable heartburn episodes
Groups:
- Vonoprazan 10 mg: On-Demand Treatment Period: Participants who had stable disease (no heartburn on the last 7 days of the Run-In Period) received oral vonoprazan 10 mg when heartburn occurred during the 6 week On-Demand Treatment Period. Participants could take no more than one dose in a 24 hour period.
- Vonoprazan 20 mg: On-Demand Treatment Period: Participants who had stable disease (no heartburn on the last 7 days of the Run-In Period) received oral vonoprazan 20 mg when heartburn occurred during the 6 week On-Demand Treatment Period. Participants could take no more than one dose in a 24 hour period.
- Vonoprazan 40 mg: On-Demand Treatment Period: Participants who had stable disease (no heartburn on the last 7 days of the Run-In Period) received oral vonoprazan 40 mg when heartburn occurred during the 6 week On-Demand Treatment Period. Participants could take no more than one dose in a 24 hour period.
- Placebo: On-Demand Treatment Period: Participants who had stable disease (no heartburn on the last 7 days of the Run-In Period) received oral placebo when heartburn occured during the 6 week On-Demand Treatment Period. Participants could take no more than one dose in a 24 hour period.
Arm/Group | Vonoprazan 10 mg: On-Demand Treatment Period | Vonoprazan 20 mg: On-Demand Treatment Period | Vonoprazan 40 mg: On-Demand Treatment Period | Placebo: On-Demand Treatment Period
Number analyzed (Participants) | 52 | 52 | 51 | 52
Number analyzed (evaluable heartburn episodes) | 359 | 327 | 323 | 370
percentage of heartburn episodes | 56.0 | 60.6 | 70.0 | 27.3
Statistical Analysis 1: Comparison: Vonoprazan 10 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p < 0.0001, Fisher Exact; Percentage difference = 28.7, 95% CI 2-sided [21.84 to 35.55]
Statistical Analysis 2: Comparison: Vonoprazan 20 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p < 0.0001, Fisher Exact; Percentage difference = 33.3, 95% CI 2-sided [26.28 to 40.23]
Statistical Analysis 3: Comparison: Vonoprazan 40 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p < 0.0001, Fisher Exact; Percentage difference = 42.7, 95% CI 2-sided [35.92 to 49.42]

2. Secondary Outcome: Percentage of Evaluable Heartburn Episodes Completely Relieved Within 3 Hours After Taking Study Drug
Description: An evaluable heartburn episode was an episode for which study drug was taken and for which the participant completed at least one entry in the heartburn episode diary.
  For a heartburn episode to be considered completely relieved, a participant must not have taken rescue antacid within 3 hours of taking study drug.
Time Frame: On-Demand Treatment Period: Day 1 to Day 42
Population: ITT On-Demand Set: includes all participants in the Safety Run-In set who were randomized and completed at least one heartburn episode diary during the On-Demand Treatment Period.
Measure: Number; unit: percentage of heartburn episodes
Units Other Than Participants: evaluable heartburn episodes
Arm/Group | Vonoprazan 10 mg: On-Demand Treatment Period | Vonoprazan 20 mg: On-Demand Treatment Period | Vonoprazan 40 mg: On-Demand Treatment Period | Placebo: On-Demand Treatment Period
Number analyzed (Participants) | 52 | 52 | 51 | 52
Number analyzed (evaluable heartburn episodes) | 359 | 327 | 323 | 370
percentage of heartburn episodes | 72.1 | 65.7 | 79.6 | 41.9
Statistical Analysis 1: Comparison: Vonoprazan 10 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p < 0.0001, Fisher Exact; Percentage difference = 30.3, 95% CI 2-sided [23.41 to 37.09]
Statistical Analysis 2: Comparison: Vonoprazan 20 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p < 0.0001, Fisher Exact; Percentage difference = 23.9, 95% CI 2-sided [16.67 to 31.05]
Statistical Analysis 3: Comparison: Vonoprazan 40 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p < 0.0001, Fisher Exact; Percentage difference = 37.7, 95% CI 2-sided [31.00 to 44.35]

3. Secondary Outcome: Percentage of Evaluable Heartburn Episodes for Each Participant That Are Completely Relieved Within 3 Hours and With No Further Heartburn Reported for 24 Hours After Taking Study Drug
Description: as for outcome 1
Time Frame: On-Demand Treatment Period: Day 1 to Day 42
Population: ITT On-Demand Set: includes all participants in the Safety Run-In set who were randomized and completed at least one heartburn episode diary during the On-Demand Treatment Period. Only participants with at least one evaluable heartburn episode during the On-Demand Treatment Period are included.
Measure: Mean (Standard Deviation); unit: % of heartburn episodes per participant
Arm/Group | Vonoprazan 10 mg: On-Demand Treatment Period | Vonoprazan 20 mg: On-Demand Treatment Period | Vonoprazan 40 mg: On-Demand Treatment Period | Placebo: On-Demand Treatment Period
Number analyzed (Participants) | 46 | 42 | 43 | 43
% of heartburn episodes per participant | 60.08 (38.452) | 60.78 (37.458) | 71.99 (28.894) | 47.77 (40.998)
Statistical Analysis 1: Comparison: Vonoprazan 10 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p = 0.1771, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Vonoprazan 20 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p = 0.1551, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Vonoprazan 40 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p = 0.0094, Wilcoxon rank-sum test

4. Secondary Outcome: Mean Number of Tablets of Rescue Antacid Taken Per Day Over the On-Demand Treatment Period
Time Frame: On-Demand Treatment Period: Day 1 to Day 42
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tablets of rescue antacid per day
Arm/Group | Vonoprazan 10 mg: On-Demand Treatment Period | Vonoprazan 20 mg: On-Demand Treatment Period | Vonoprazan 40 mg: On-Demand Treatment Period | Placebo: On-Demand Treatment Period
Number analyzed (Participants) | 52 | 52 | 51 | 52
tablets of rescue antacid per day | 0.1 (0.21) | 0.2 (0.29) | 0.1 (0.26) | 0.5 (0.87)
Statistical Analysis 1: Comparison: Vonoprazan 10 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p = 0.3395, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Vonoprazan 20 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p = 0.4882, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Vonoprazan 40 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p = 0.0722, Wilcoxon rank-sum test

5. Secondary Outcome: Percentage of Participants With Complete Relief of Heartburn Within 3 Hours After the First Episode and With No Further Heartburn Reported for 24 Hours After Taking Study Drug
Description: as for outcome 1
Time Frame: On-Demand Treatment Period: Day 1 to Day 42
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Vonoprazan 10 mg: On-Demand Treatment Period | Vonoprazan 20 mg: On-Demand Treatment Period | Vonoprazan 40 mg: On-Demand Treatment Period | Placebo: On-Demand Treatment Period
Number analyzed (Participants) | 46 | 42 | 43 | 43
percentage of participants | 56.5 | 61.9 | 62.8 | 60.5
Statistical Analysis 1: Comparison: Vonoprazan 10 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p = 0.8300, Fisher Exact; Percentage difference = -3.9, 95% CI 2-sided [-24.41 to 16.52]
Statistical Analysis 2: Comparison: Vonoprazan 20 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p > 0.9999, Fisher Exact; Percentage difference = 1.4, 95% CI 2-sided [-19.28 to 22.16]
Statistical Analysis 3: Comparison: Vonoprazan 40 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p > 0.9999, Fisher Exact; Percentage difference = 2.3, 95% CI 2-sided [-18.22 to 22.88]

6. Secondary Outcome: Percentage of Days Study Drug Was Taken Over the On-Demand Treatment Period
Time Frame: On-Demand Treatment Period: Day 1 to Day 42
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Vonoprazan 10 mg: On-Demand Treatment Period | Vonoprazan 20 mg: On-Demand Treatment Period | Vonoprazan 40 mg: On-Demand Treatment Period | Placebo: On-Demand Treatment Period
Number analyzed (Participants) | 52 | 52 | 51 | 52
percentage of days | 21.93 (19.241) | 20.75 (16.950) | 21.01 (17.302) | 22.15 (23.266)
Statistical Analysis 1: Comparison: Vonoprazan 10 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p = 0.4684, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Vonoprazan 20 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p = 0.6560, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Vonoprazan 40 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p = 0.6324, Wilcoxon rank-sum test

7. Secondary Outcome: Percentage of 24-Hour Heartburn-Free Days Over the On-Demand Treatment Period
Description: A 24-hour heartburn-free day was defined as a day having no heartburn among all diary entries for that day. The percentage of 24-hour heartburn-free days was calculated using all days with at least 1 evening or morning diary entry during the treatment period of this phase.
Time Frame: On-Demand Treatment Period: Day 1 to Day 42
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Vonoprazan 10 mg: On-Demand Treatment Period | Vonoprazan 20 mg: On-Demand Treatment Period | Vonoprazan 40 mg: On-Demand Treatment Period | Placebo: On-Demand Treatment Period
Number analyzed (Participants) | 52 | 52 | 51 | 52
percentage of days | 74.95 (21.410) | 73.57 (21.465) | 74.01 (22.277) | 71.22 (28.867)
Statistical Analysis 1: Comparison: Vonoprazan 10 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p = 0.9896, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Vonoprazan 20 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p = 0.6916, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Vonoprazan 40 mg: On-Demand Treatment Period vs Placebo: On-Demand Treatment Period; Test type: Superiority; p = 0.9316, Wilcoxon rank-sum test

ADVERSE EVENTS:
Time Frame: Run-In Period: Day 1 to Day 28; On-Demand Treatment: Day 1 to Day 49
Description: Run-In Period: The Safety Run-In Set includes participants who received at least one dose of vonoprazan during the Run-In Period.
  On-Demand Treatment Period: The Safety On Demand Set includes all participants in the Safety Run-In Set who were randomized and treated at least one heartburn episode with randomized treatment during the On-Demand Treatment period.
Groups:
- Run-In Period: Participants received oral vonoprazan 20 mg QD for up to 4 weeks.
Arm/Group | Run-In Period | Vonoprazan 10 mg: On-Demand Treatment Period | Vonoprazan 20 mg: On-Demand Treatment Period | Vonoprazan 40 mg: On-Demand Treatment Period | Placebo: On-Demand Treatment Period
All-Cause Mortality (participants affected / at risk) | 0/457 | 0/49 | 0/49 | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 4/457 | 0/49 | 0/49 | 0/48 | 0/47
Other Adverse Events (participants affected / at risk) | 29/457 | 8/49 | 9/49 | 8/48 | 10/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In Period (N=457) | Vonoprazan 10 mg: On-Demand Treatment Period (N=49) | Vonoprazan 20 mg: On-Demand Treatment Period (N=49) | Vonoprazan 40 mg: On-Demand Treatment Period (N=48) | Placebo: On-Demand Treatment Period (N=47)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In Period (N=457) | Vonoprazan 10 mg: On-Demand Treatment Period (N=49) | Vonoprazan 20 mg: On-Demand Treatment Period (N=49) | Vonoprazan 40 mg: On-Demand Treatment Period (N=48) | Placebo: On-Demand Treatment Period (N=47)
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 6 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 4 | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 2 | 1 | 1 | 1 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 3 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 1 | 0 | 0 | 0
Urine analysis abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 1 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT04799158/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT04799158/SAP_001.pdf